CLINICAL TRIAL: NCT07161232
Title: The Influence of the Timing of Postoperative Rehabilitation Intervention on the Clinical
Brief Title: The Influence of the Timing of Postoperative Rehabilitation Intervention on the Clinical Efficacy of Unilateral Biportal Endoscopic Spine System in the Treatment of Lumbar Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Li Xiang (Other)
Responsible Party: Sponsor-Investigator, Li Xiang, chief physician, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-P2-070-02
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Disc Herniation; Postoperative Rehabilitation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Rehabilitation Group (Experimental): Patients in this arm will commence a standardized, progressive rehabilitation program at 2 weeks (±3 days) following unilateral biportal endoscopic (UBE) surgery. The regimen consists of core stability exercises and neurodynamic techniques designed to early activate core muscles, prevent neural adhesion, and restore function. Specific exercises include transverse abdominis activation, sit-to-stand training with abdominal bracing, four-point kneeling rockbacks for spinal mobility, neural mobilization in the modified straight leg raise position, and neural sliding techniques. The exercises are performed once daily and progressed based on patient tolerance. The entire intervention is supervised by a senior physical therapist.
  Interventions: Behavioral: Standardized Postoperative Rehabilitation Protocol
- Late Rehabilitation Group (Active Comparator): This arm serves as the active comparator. Patients will commence the identical standardized, progressive rehabilitation program as the Experimental arm at 6 weeks (±3 days) following unilateral biportal endoscopic (UBE) surgery. The content of the rehabilitation regimen, exercise frequency, progression criteria, and supervision by a physical therapist are exactly the same as in the Experimental arm. This timing represents the conventional, later postoperative rehabilitation approach.
  Interventions: Behavioral: Standardized Postoperative Rehabilitation Protocol

INTERVENTIONS:
Behavioral: Standardized Postoperative Rehabilitation Protocol — This intervention is a standardized, progressive rehabilitation protocol for patients after lumbar disc herniation surgery, delivered under the guidance of a senior physical therapist. The protocol aims to improve pain, restore function, and prevent complications through core stability exercises and neurodynamic techniques. The exercises are performed once daily and progressed based on patient tolerance. The protocol consists of two phases:
  Initial Phase ( commencing postoperatively): Includes: 1) Transverse abdominis activation; 2) Sit-to-stand training with abdominal bracing; 3) Four-point kneeling rockbacks for spinal mobility; 4) Neural mobilization techniques (performed in sitting); 5) Neural sliding techniques (performed in sitting).
  Progressive Phase: Builds upon the initial exercises by increasing the range of motion, adding isometric hold times, and integrating cervical movement with neural techniques to increase difficulty and intensity.

SUMMARY:
This study focuses on the impact of the timing of postoperative rehabilitation intervention on the clinical efficacy of unilateral biportal endoscopic spine surgery in the treatment of lumbar disc herniation. The main objective is to explore this impact and provide high-quality evidence-based medical evidence for making reasonable clinical decisions.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial on the impact of the timing of postoperative rehabilitation intervention on the clinical efficacy of unilateral biportal endoscopic spine surgery in the treatment of lumbar disc herniation. The main purpose is to explore this impact and provide high-quality evidence-based medical evidence for making reasonable clinical decisions. According to the inclusion and exclusion criteria formulated in this study, 72 patients who underwent UBE surgery for lumbar disc herniation were recruited in our hospital and randomly assigned to the early rehabilitation intervention group (referred to as the early rehabilitation group, with rehabilitation intervention starting 2 weeks after surgery) or the late rehabilitation intervention group (referred to as the late rehabilitation group, with rehabilitation intervention starting 6 weeks after surgery) after surgery. The clinical and subjective (questionnaire) data of the subjects before surgery, after surgery and during the follow-up process (up to 12 months after surgery) were collected to compare the differences in clinical efficacy between early and late postoperative rehabilitation intervention in patients with lumbar disc herniation treated by UBE.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 65 years.

Diagnosed with lumbar disc herniation by imaging and scheduled for unilateral biportal endoscopic (UBE) surgery.

Presenting with radicular pain in the lower extremity, with a history of less than 1 year.

Able to understand Chinese and complete questionnaires independently.

Physically capable of participating in exercise rehabilitation.

Willing to participate and provide written informed consent.

Exclusion Criteria:

* Aged under 18 or over 65 years.

Combined with other spinal pathologies (e.g., ankylosing spondylitis, rheumatoid arthritis, spinal tumor, spinal fracture, cauda equina syndrome).

Diagnosis of neurological disorders (e.g., multiple sclerosis, Parkinson's disease).

Presence of uncontrolled cardiovascular, respiratory, or peripheral vascular diseases.

History of severe psychiatric disorders (e.g., schizophrenia).

Previous history of spinal surgery.

Pregnancy or lactation.

Inability to understand or comply with the study procedures.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Score | Change from Baseline to 12 months postoperatively
  The Oswestry Disability Index (ODI) is a widely validated and disease-specific patient-reported outcome measure for assessing functional status in individuals with low back pain. The questionnaire consists of 10 items addressing pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment/homemaking. Each item is scored from 0 to 5, and the total score is converted to a percentage (0-100%), with higher scores indicating greater disability. The ODI score at 12 months postoperatively will be used as the primary endpoint to evaluate the long-term effect of rehabilitation timing.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The ethical approval and patient informed consent forms obtained for this study are applicable only for the current research objectives and do not include provisions for public sharing of individual data. To protect patient privacy and comply with ethical regulations, we are unable to publicly share IPD at this time.